CLINICAL TRIAL: NCT05953051
Title: A Single-center, Patient-blinded, Randomized, 2-year, Parallel-group, Superiority Study to Compare the Efficacy of Augmented ACL Integration Via Platelet-rich-plasma Enriched Collected Autologous Bone Versus Standard ACL Technique
Brief Title: Tunnel Widening in Augmented ACL Integration Via PrP Enriched Collected Autologous Bone vs Standard ACL Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UE-0073; 2022-00168 (Other: BASEC)
Record Dates: First submitted 2023-06-29; First posted 2023-07-19 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: Anterior Cruciate Ligament Reconstruction; Platelet-Rich Plasma; Bone Tunnel Widening
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Patients will be allocated 1:1 on experimental and control arm using block randomization within both genders with random block sizes (randomly chosen from the set [2,4,6,8]).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are blinded. As well, staff conducting and evaluating MRI, clinical evaluation, CT and functional tests are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACLr with bone/PrP-composite (Experimental): During surgery, the drilled bone debris is collected in a sterile filtered chamber.
  Then the bone debris is mixed with PrP. After fixation of the graft the composite is inserted into the drilled tunnel at the interface between tendon to bone. The intraarticular aperture sites are sealed by use of fibrin that is previously gathered out of the PrP as well.
  Interventions: Procedure: ACL reconstruction with bone/PrP-composite
- ACLr standard (Active Comparator): No insertion of additional material after ACL graft fixation.
  Interventions: Procedure: ACL reconstruction (Standard)

INTERVENTIONS:
Procedure: ACL reconstruction with bone/PrP-composite — During standard ACL reconstruction, the drilled bone debris is collected in a sterile filtered chamber.
  Then the bone debris is mixed with PrP. After fixation of the graft the composite is inserted into the drilled tunnel at the interface between tendon to bone. The intraarticular aperture sites are sealed by use of fibrin that is previously gathered out of the PrP as well.
  Arms: ACLr with bone/PrP-composite
Procedure: ACL reconstruction (Standard) — Standard ACL reconstruction with Semitendinosus alone or plus gracilis, femoral fixation via extracortical fixation by adjustable loop device, tibial fixation via a bio-interference screw or adjustable device
  Arms: ACLr standard

SUMMARY:
The purpose of this clinical study is to compare the outcomes of two surgical techniques for reconstruction of the anterior cruciate ligament (ACL) after a single, primary ACL rupture.

The main question to be answered is:

- Does less widening of the tibial tunnel occur when a bone/Platelet rich plasma (PrP) composite material is placed directly into the tibial tunnel after fixation of the implant (experimental group) compared to the same surgery without the use of the composite material (control group)?

Participants will be randomized into one of the two groups and they will not know which group they belong to. After 12 months they will undergo CT, MRI, medical examination and functional knee testing. They will have a further medical examination and functional knee testing at 24 months. Patient Reported Outcomes will be collected before surgery, 6, 12 and 24 months after surgery.

DETAILED DESCRIPTION:
To be successful, an ACL reconstruction requires a strong incorporation of the tendon to the bone within or at the margin of the tunnel, but the tunnel itself is at risk of widening, therefore compromising the tendon attachment. A composite of harvested healthy autologous bone fragments from the tunnel and autologous thrombin and fibrin, generated from the patient's PrP could be used at the interface between tunnel and ACL graft at the tibia and femur to reduce frequency of tunnel widening and therefore improve graft-bone-integration.

The study seeks primarily to determine less tibial tunnel widening when a bone/PrP-composite is applied directly in the tibial tunnel compared to the same surgery without using the composite, measured with CT and MRI.

Secondary study objectives are to evaluate femoral tunnel widening, tibial and femoral graft incorporation, graft maturation and knee function (clinical, functional, patient reported) over the course of 24 months follow-up and to evaluate occurrence of procedure- and product-related adverse events and complications.

This is a prospective, single-center, single-blinded, 2-arm-parallel, randomized, controlled study with 24 months follow-up. Participants will be recruited from the Knee Surgery department at Schulthess Klinik when scheduled for ACL reconstruction. The study sample comprises 107 patients, allocated 1:1 on experimental and control arm. Outcome measures are taken at 0, 6, 12, and 24 months. The total study duration is 48 months. The study duration per patient is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Primary ACL rupture
* Time from injury to surgery: 4 weeks to 6 months
* Single ACL rupture (isolated rupture)
* ACL surgery with one of the participating senior surgeons
* Informed Consent as documented by signature

Exclusion Criteria:

* Concomitant ligamentous instability/rupture
* Requirement for Meniscus suture (partial resection accepted, hoop and roots remain intact)
* Requirement for cartilage invasive treatment (debridement accepted)
* Osteoarthritis at index knee joint
* Leg axis deviation over 3° valgus or 4° varus
* Claustrophobia (contra-indication for the MRI)
* Women who are pregnant or breast feeding or intention to become pregnant during the study
* Known or suspected non-compliance, drug or alcohol abuse
* Inability of the patient to follow the study procedures, e.g. language problems, psychological disorders, dementia, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Tibial tunnel diameter change | 10 to 14 months post-surgery
  Diameter (mm) change of tibial tunnel in relation to tunnel diameter reported from surgery; assessed by one radiologist (CT); CT scanning is performed from a level just above the femoral external foramen to a level below the outer hole of the tibial tunnel in order to visualise the positioning of the autograft-fixing metallic devices. The scan is aligned so that the tunnel axis is in the sagittal plane. The diameter of the headed reamer that drilled the tibial tunnel is defined as the baseline diameter of the tibial tunnel (D0). Measurements are taken at 4 different levels for the tibial tunnels using 3D Multiplanar reconstruction. All diameters are calculated in mm within the measurement function of the picture archiving system. The percentage of widening is defined as the difference between initial drilling diameter D0 (derived from surgery report) and post-op measurements D12 in relation to initial drilling diameter D0.
Tibial tunnel volume change | 10 to 14 months post-surgery
  Volume (mm^3) change of tibial tunnel in relation to tunnel volume reported from surgery; assessed by one radiologist (CT); the border of the bone tunnel is drawn manually on every fourth slice in both the coronal plane and the sagittal plane and interpolated automatically in between. Based on the contours in those two planes, the contours in the axial plane are interpolated automatically into a 3D mask. The volume of the bone tunnel is determined by automatic voxel counting^.

SECONDARY OUTCOMES:
Femoral tunnel diameter change | 10 to 14 months post-surgery
  Diameter (mm) change of femoral tunnel in relation to tunnel diameter reported from surgery; assessed by one radiologist (CT); CT scanning is performed from a level just above the femoral external foramen to a level below the outer hole of the tibial tunnel in order to visualise the positioning of the autograft-fixing metallic devices. The scan is aligned so that the tunnel axis is in the sagittal plane. The diameter of the headed reamer that drilled the femoral tunnel is defined as the baseline diameter of the femoral tunnel (D0). Measurements are taken at 4 different levels for the femoral tunnels using 3D Multiplanar reconstruction. All diameters are calculated in mm within the measurement function of the picture archiving system. The percentage of widening is defined as the difference between initial drilling diameter D0 (derived from surgery report) and post-op measurements D12 in relation to initial drilling diameter D0.
Femoral tunnel volume change | 10 to 14 months post-surgery
  Volume (mm^3) change of femoral tunnel in relation to tunnel volume reported from surgery; assessed by one radiologist (CT); the border of the bone tunnel is drawn manually on every fourth slice in both the coronal plane and the sagittal plane and interpolated automatically in between. Based on the contours in those two planes, the contours in the axial plane are interpolated automatically into a 3D mask. The volume of the bone tunnel is determined by automatic voxel counting.
Graft maturity_subj | 10 to 14 months post-surgery
  tibial & femoral, subjectively, using a 4-grade system MRI after 12 months based on Proton-density-weighted images
  * Grade 1 signal ("normal"): when the entire segment of graft has a homogeneous, low intensity signal indistinguishable from that of the posterior cruciate ligament
  * Grade 2: if the segment of graft retained at least 50% of "normal" ligament signal intermixed with portions of the graft that had become edematous, as indicated by areas of increased signal intensity
  * Grade 3: when a segment of graft had ~50% of its area exhibiting a normal appearing ligament signal
  * Grade 4: diffuse increase in signal intensity with no normal-looking strands of ligament (100% oedematous).
Graft maturity_obj | 10 to 14 months post-surgery
  objectively, within the tibial and femoral tunnels and in the intra-articular portion using the mean intensity of a region of interest on MRI to estimate the graft signal to noise quotient (SNQ) in comparison to the quadriceps tendon: SNQ = Signal intensity graft - Signal intensity quadriceps tendon / SI background
Graft integration | 10 to 14 months post-surgery
  tibial & femoral,
  * Grade I, full attachment of a low-intensity signal band onto the bone tunnel with no fibrous tissue at the tendon-bone interface;
  * Grade II, a low-intensity signal band with a partial high- intensity signal band at the tendon-bone interface;
  * Grade III, the graft bone interface is filled with a continuous high- intensity signal band.
Bone healing and integration | 10 to 14 months post-surgery
  subjectively, tibial & femoral, of the applied autologous bone matrix
  * Grade I, excellent integration indicating no space between the graft and osseous formation in the proximal and mid portion.
  * Grade II, good integration indicating no space between the graft and osseous formation in the proximal or mid portion.
  * Grade III, fair integration indicating a gap between the graft and osseous formation in the proximal and mid portion.
  * Grade IV, poor integration indicating no osseous formation in the proximal and mid portion.

OTHER OUTCOMES:
Range of motion | 10-14 and 20-28 months post-surgery
  extension and flexion (°) both knees
Isokinetic knee strength test | 10-14 and 20-28 months post-surgery
  Extension and Flexion (Nm), operated vs. non-operated side
Y-balance test | 10-14 and 20-28 months post-surgery
  balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial
Knee Laxity | 10-14 and 20-28 months post-surgery
  the patient is placed in the supine position on an examination table, the knees remain at approximately 30° of flexion and the tibia a 15° rotation. The displacement is consequently measured with the KT-1000 arthrometer device, calculating the relative motion between the sensor pad on the patella and the sensor pad on the anterior tibia under 67, 89 and 134 N force. The healthy leg is always to be tested first followed by the injured leg. The side-to-side differences are then evaluated at each force (mm)
Front hop | 10-14 and 20-28 months post-surgery
  unilateral forward jump as far as possible (cm)
Side hop | 10-14 and 20-28 months post-surgery
  repeated side hops over a distance of 40 cm and back to start position (number of touch-downs within 30 seconds)
gait restrictions | 10-14 and 20-28 months post-surgery
  gait restrictions related to the operated knee (i.e. limping) (y/n)
adverse events | 10-14 and 20-28 months post-surgery
  procedure- and product-related adverse events will be described and given as frequency per type
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | -3 to 0, 6, 12, 24 months post-surgery
  standardized instrument for measuring generic health status regardless of existing diseases within five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), result is a 5-level health state
EuroQol visual analogue scale (EQ-VAS) | -3 to 0, 6, 12, 24 months post-surgery
  Quality of life, regardless of existing diseases, visual analogue scale from 0 - 100. 0 points correspond to the worst possible health status, while 100 points correspond to the best possible health status.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | -3 to 0, 6, 12, 24 months post-surgery
  assess patient-relevant outcomes following knee injury using 42 items within 5 subscales, which are scored separately; each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Tegner Activity Scale | 12, 24 months post-surgery
  one-item score that grades activity based on work and sports activities on a scale of 0 (disability because of knee problems) to 10 (national or international elite level)
Return to Sport Injury Scale (ACL-RSI) | 12, 24 months post-surgery
  the patient's self-confidence and risk assessment regarding a return to sport after ACL reconstruction with 12 items using a numeric rating scale of 0 to 100.
Numeric Rating scale for pain (NRS) in the knee | -3 to 0, 6, 12, 24 months post-surgery
  unidimensional measure of pain intensity in adults, where 0=no pain and 10=worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Gian Salzmann, Prof., Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
When published, authors will make their data available upon reasonable request or according to the guidelines of the journal.